CLINICAL TRIAL: NCT00865189
Title: Efficacy and Safety of Two Neoadjuvant Strategies With Bevacizumab in Locally Advanced Resectable Rectal Cancer: A Randomized, Non-Comparative Phase II Study
Brief Title: A Study of Bevacizumab (Avastin) in Participants With Newly Diagnosed Locally Advanced Rectal Cancer
Acronym: INOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19202; 2006-003472-35 (EudraCT Number)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil; Surgical Procedures, Operative

ARMS (2):
- Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) (Experimental): In this arm, participants will undergo 3 phases of treatment. During the Phase 1, participants will receive induction chemotherapy with 6 two-week cycles of bevacizumab + Folfox-4 (5-FU + oxaliplatin + folinic acid) for 12 weeks followed by a treatment-free interval of 3 to 4 weeks. The Phase 2 will include 7 weeks of bevacizumab + chemoradiotherapy (intravenous [IV] infusion of bevacizumab alone, 2 weeks before administration of the first cycle of chemoradiotherapy, then 5 one-week cycles of chemoradiotherapy [5-FU + radiotherapy], with administration of bevacizumab every two weeks [Cycles 1, 3 and 5]) followed by a treatment-free interval of 6 to 8 weeks. The Phase 3 will be surgery involving a radical rectal excision using the total mesorectal excision (TME) technique.
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluorouracil; Radiation: Preoperative Radiotherapy; Procedure: Surgery
- Arm B (Bevacizumab, Chemoradiotherapy) (Experimental): In this arm, participants will receive the Phase 2 and Phase 3 treatments only. The phase 2 will include 7 weeks of bevacizumab + chemoradiotherapy (IV infusion of bevacizumab alone, 2 weeks before administration of the first cycle of chemoradiotherapy, then 5 one-week cycles of chemoradiotherapy [5-FU + radiotherapy], with administration of bevacizumab every two weeks [Cycles 1, 3 and 5]) followed by a treatment-free interval of 6 to 8 weeks. The phase 3 will be surgery involving a radical rectal excision using the TME technique.
  Interventions: Drug: Bevacizumab; Drug: 5-fluorouracil; Radiation: Preoperative Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at the fixed dose of 5 milligrams per kilogram (mg/kg) as an IV infusion over 30 to 90 minutes.
  Other Names: Avastin
Drug: Oxaliplatin — Oxaliplatin will be administered at a dose of 85 milligrams per square meter (mg/m^2) as a 2-hour IV infusion.
  Arms: Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy)
Drug: Folinic Acid — Folinic acid will be administered at a dose of 200 mg/m^2 as a 2-hour infusion.
  Arms: Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy)
Drug: 5-fluorouracil — 5-fluorouracil will be administered at a dose of 400 mg/m^2 as an IV bolus, then at a dose of 600 mg/m^2 as a continuous infusion for 22 hours in Phase 1, and will be administered at a dose of 225 mg/m^2 as a 24-hour infusion, 5 days a week, for 5 weeks in Phase 2.
Radiation: Preoperative Radiotherapy — Radiotherapy will be delivered in fraction of 1.8 gray per day (Gy/day), 5 days a week for 5 weeks, i.e., a total dose of 45 Gy will be administered in 25 fractions over a period of 33 days.
Procedure: Surgery — Radical rectal excision based on the TME technique.

SUMMARY:
This study will assess the efficacy and safety of two different neoadjuvant treatment approaches including bevacizumab in newly diagnosed participants with high risk locally advanced rectal cancer. Participants will be randomized into one of two treatment arms (Arm A or Arm B).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed locally advanced rectal cancer;
* measurable disease;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Exclusion Criteria:

* prior treatment with bevacizumab;
* prior radiotherapy to pelvic region, or previous cytotoxic chemotherapy;
* previous history of malignancy (other than basal and squamous cell cancer of the skin, or in situ cancer of the cervix);
* history or evidence of central nervous system (CNS) disease;
* clinically significant cardiovascular disease;
* chronic treatment with high dose aspirin (more than [>] 325 milligrams per day [mg/day]) or non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-10-23 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (38):
- France (38):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Angers
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Besançon
  - Hopital Saint Andre; Département de Radiothérapie Et D'Oncologie Médicale, Bordeaux
  - Bordeaux
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Dijon
  - Hopital Albert Michallon; Radiotherapie, La Tronche
  - La Tronche
  - Centre Oscar Lambret; Radiotherapie, Lille
  - Lille
  - Centre Hospitalier Andre Boulloche; Departement D'Oncologie, Montbéliard
  - Montbéliard
  - Centre Val Aurelle Paul Lamarque; Radiotherapie, Montpellier
  - Montpellier
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Nancy
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Nice
  - Hopital Saint Louis; Radiotherapie Oncologie, Paris
  - Paris
  - Ch Pitie Salpetriere; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Ch Lyon Sud; Radiotherapie Sct Jules Courmont, Pierre-Bénite
  - Pierre-Bénite
  - Chu La Miletrie; Radiotherapie, Poitiers
  - Poitiers
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Saint-Herblain
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Strasbourg
  - Polyclinique Du Parc; Centre De Hautes Energies, Toulouse
  - Toulouse
  - Hopital Bretonneau; Clinique D'Oncologie & de Radiotherapie, Tours
  - Tours
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Borg C, Andre T, Mantion G, Boudghene F, Mornex F, Maingon P, Adenis A, Azria D, Piutti M, Morsli O, Bosset JF. Pathological response and safety of two neoadjuvant strategies with bevacizumab in MRI-defined locally advanced T3 resectable rectal cancer: a randomized, noncomparative phase II study. Ann Oncol. 2014 Nov;25(11):2205-2210. doi: 10.1093/annonc/mdu377. Epub 2014 Aug 13. PMID 25122693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 92 participants with resectable rectal cancer were selected and 91 participants were randomized into the study. One participant was not randomized due to non-compliance with the inclusion/exclusion criteria.
Groups:
- Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy): In this arm, participants underwent 3 phases of treatment. During the Phase 1, participants received induction chemotherapy with 6 two-week cycles of bevacizumab + Folfox-4 (5-FU + oxaliplatin + folinic acid) for 12 weeks followed by a treatment-free interval of 3 to 4 weeks. The Phase 2 consisted of 7 weeks of bevacizumab + chemoradiotherapy (intravenous [IV] infusion of bevacizumab alone, 2 weeks before administration of the first cycle of chemoradiotherapy, then 5 one-week cycles of chemoradiotherapy [5-FU + radiotherapy], with administration of bevacizumab every two weeks [Cycles 1, 3 and 5]) followed by a treatment-free interval of 6 to 8 weeks. The Phase 3 was surgery involving a radical rectal excision using the total mesorectal excision (TME) technique.
- Arm B (Bevacizumab, Chemoradiotherapy): In this arm, participants received the Phase 2 and Phase 3 treatments only. The phase 2 consisted of 7 weeks of bevacizumab + chemoradiotherapy (IV infusion of bevacizumab alone, 2 weeks before administration of the first cycle of chemoradiotherapy, then 5 one-week cycles of chemoradiotherapy [5-FU + radiotherapy], with administration of bevacizumab every two weeks [Cycles 1, 3 and 5]) followed by a treatment-free interval of 6 to 8 weeks. The phase 3 was surgery involving a radical rectal excision using the TME technique.
Period: Overall Study
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Started | 46 | 45
Completed | 34 | 26
Not Completed | 12 | 19
Not completed — Other | 1 | 2
Not completed — Death | 4 | 11
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all the randomized participants who received at least one dose of treatment.
Groups:
- Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy): In this arm, participants underwent 3 phases of treatment. During the Phase 1, participants received induction chemotherapy with 6 two-week cycles of bevacizumab + Folfox-4 (5-FU + oxaliplatin + folinic acid) for 12 weeks followed by a treatment-free interval of 3 to 4 weeks. The Phase 2 consisted of 7 weeks of bevacizumab + chemoradiotherapy (IV infusion of bevacizumab alone, 2 weeks before administration of the first cycle of chemoradiotherapy, then 5 one-week cycles of chemoradiotherapy [5-FU + radiotherapy], with administration of bevacizumab every two weeks [Cycles 1, 3 and 5]) followed by a treatment-free interval of 6 to 8 weeks. The Phase 3 was surgery involving a radical rectal excision using the TME technique.
- Total: Total of all reporting groups
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy) | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 29 | 62
  >=65 years | 13 | 16 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tumor Sterilization Defined by ypT0-N0
Description: Tumor sterilization was defined as the absence of residual tumor cells in the resected specimen including lymph nodes (ypT0-N0). The rate of sterilization of the tumoral specimen was assessed after surgery on the surgical specimen by local review. Analyses were performed for participants who have been operated as defined by the protocol (within the study and TME technique) and for all participants who have been operated. Reported is the percentage of participants with tumor sterilization.
Time Frame: After surgery (Arm A: approximately 28-31 weeks after initiation of treatment; Arm B: approximately 13-15 weeks after initiation of treatment)
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 42 | 44
percentage of participants | 23.8 [12.1 to 39.5] | 11.4 [3.8 to 24.6]
Statistical Analysis 1: Comparison: Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy); This proportion was described for each treatment arm with a 95% confidence interval (CI) and compared with the standard proportion of 10% (CI) for each treatment arm; Test type: Superiority or Other; p = 0.015, Binomial test
Statistical Analysis 2: Comparison: Arm B (Bevacizumab, Chemoradiotherapy); This proportion was described for each treatment arm with a 95% CI and compared with the standard proportion of 10% (CI) using for each treatment arm; Test type: Superiority or Other; p = 0.906, Binomial test

2. Secondary Outcome: Percentage of Participants With Tumor Down-Staging (ypT0-pT2)
Description: A participant with a downstaging was defined as a participant with T3 (T describes the size of the original [primary] tumor) at inclusion and T2 or T1 or T0 after surgery, or with N+ (N describes lymph nodes involvement) at inclusion and N- after surgery and if T is equal at inclusion and after surgery. The clinical tumor-node-metastasis (cTNM) classification was used at inclusion and the pathological staging tumor and nodes (ypTN) classification after surgery. Reported is the percentage of participants with tumor downstaging of the surgical specimen according to the local review and centralized review.
Time Frame: as for outcome 1
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome. "n" = participants who were evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 41 | 44
percentage of participants
  Downstaging, local review (n=41, 44) | 65.9 [51.3 to 80.4] | 54.5 [39.8 to 69.3]
  Downstaging, centralized review (n=39, 43) | 64.1 [49.0 to 79.2] | 55.8 [41.0 to 70.7]

3. Secondary Outcome: Percentage of Participants With Local and Distant Recurrences
Description: The percentage of participants with a recurrence was described by type of recurrence (local and distant recurrence).
Time Frame: as for outcome 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
percentage of participants
  Local recurrence | 2.2 [0.1 to 11.5] | 6.7 [1.4 to 18.3]
  Distant recurrence | 17.4 [7.8 to 31.4] | 13.3 [5.1 to 26.8]

4. Secondary Outcome: Percentage of Participants With Second Cancer, Local or Regional Recurrence, Distant Metastasis, or Death
Time Frame: Baseline up to approximately 6 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
percentage of participants | 30.4 [1.4 to 18.3] | 33.3

5. Secondary Outcome: Disease-Free Survival (DFS)
Description: The DFS was defined as the time from the first treatment intake to disease recurrence assessed (second primary cancer, local or distant recurrence, distant metastases) or death from any cause. The DFS was analyzed using Kaplan-Meier method.
Time Frame: From first time of the treatment administration to the date of second cancer, local or regional recurrence, distant metastasis or death from any cause (up to approximately 6 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
months | 68.3 [68.3 to NA] — Upper limit of 95% CI was not reached due to low number of DFS-events. | NA [53.0 to NA] — Median and upper limit of 95% CI were not reached due to low number of DFS-events.

6. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline up to approximately 6 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
percentage of participants | 8.7 [1.4 to 18.3] | 24.4

7. Secondary Outcome: Overall Survival
Description: The overall survival was defined as the time from the first treatment intake to death from any cause.
Time Frame: From the first treatment administration to the date of death (up to approximately 6 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
months | NA [NA to NA] — Median and 95% CI were not reached due to low number of deaths. | NA [NA to NA] — Median and 95% CI were not reached due to low number of deaths.

8. Secondary Outcome: Number of Cycles of Induction Chemotherapy
Time Frame: 6 cycles (12 weeks; cycle length = 14 days)
Population: ITT population. Only Arm A participants received induction treatment.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy)
Number analyzed (Participants) | 46
cycles | 5.8 (0.7)

9. Secondary Outcome: Number of Cycles of Chemotherapy
Time Frame: Arm A: Week 16 to Week 23; Arm B: Week 1 to Week 7
Population: ITT population
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
cycles | 4.4 (1.5) | 4.8 (0.5)

10. Secondary Outcome: Number of Cycles of Radiotherapy
Time Frame: Arm A: Week 16 to Week 23; Arm B: Week 1 to Week 7
Population: ITT population
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
cycles | 4.5 (1.5) | 5.0 (0.0)

11. Secondary Outcome: Percentage of Participants With Surgery
Description: The surgery involving a radical rectal excision using the TME technique.
Time Frame: Arm A: approximately 28-31 weeks after initiation of treatment; Arm B: approximately 13-15 weeks after initiation of treatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Number analyzed (Participants) | 46 | 45
percentage of participants | 91.3 (0.0) | 97.8

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 6 years
Description: The safety population included all selected participants who received at least one dose of treatment and corresponded to the ITT population.
Arm/Group | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) | Arm B (Bevacizumab, Chemoradiotherapy)
Serious Adverse Events (participants affected / at risk) | 21/46 | 18/45
Other Adverse Events (participants affected / at risk) | 46/46 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) (N=46) | Arm B (Bevacizumab, Chemoradiotherapy) (N=45)
Anastomotic fistula (Injury, poisoning and procedural complications) | 4 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 2
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 2 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 2
Catheter site infection (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural infection (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Rectoprostatic fistula (Reproductive system and breast disorders) | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 1
Embolism venous (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Wernicke's encephalopathy (Nervous system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Bevacizumab, Induction Chemotherapy, Chemoradiotherapy) (N=46) | Arm B (Bevacizumab, Chemoradiotherapy) (N=45)
Diarrhoea (Gastrointestinal disorders) | 25 | 24
Nausea (Gastrointestinal disorders) | 24 | 7
Constipation (Gastrointestinal disorders) | 15 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4
Anorectal discomfort (Gastrointestinal disorders) | 1 | 7
Proctalgia (Gastrointestinal disorders) | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 6 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3
Gingivitis (Gastrointestinal disorders) | 3 | 0
Proteinuria (Renal and urinary disorders) | 20 | 13
Dysuria (Renal and urinary disorders) | 12 | 10
Pollakiuria (Renal and urinary disorders) | 2 | 3
Asthenia (General disorders) | 17 | 6
Mucosal inflammation (General disorders) | 7 | 4
Fatigue (General disorders) | 4 | 2
Pyrexia (General disorders) | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 22 | 0
Paraesthesia (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 7 | 2
Dysaesthesia (Nervous system disorders) | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 5
Anastomotic fistula (Injury, poisoning and procedural complications) | 3 | 2
Wound complication (Injury, poisoning and procedural complications) | 4 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 3 | 1
Neutrophil count decreased (Investigations) | 12 | 1
Blood potassium decreased (Investigations) | 5 | 1
Weight decreased (Investigations) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 11 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Proctitis (Gastrointestinal disorders) | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.